CLINICAL TRIAL: NCT07373184
Title: Three-dimensional Virtual Planning of Total Temporomandibular Joint Replacement Using Standardized Prosthesis.
Brief Title: Virtual Planning of Total Temporomandibular Joint Replacement
Status: Recruiting | Type: Observational
Sponsor: Lund University Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-01826-01
Record Dates: First submitted 2025-12-11; First posted 2026-01-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Temporomandibular Disorders (TMD); Temporomandibular Joint Ankylosis
Keywords: temporomandibular joint; temporomandibular disorder; ankylosis; joint prosthesis; total joint replacement
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular ankylosis; Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A total TMJ replacement surgery is currently planned based on the X-ray appearance of the facial X-ray. It is now possible to use either an individually designed TMJ prosthesis or a prosthesis with a standard appearance. It is a significantly higher cost for treatment with an individually manufactured prosthesis, but it also provides the opportunity for virtual planning of the positioning of the jaws and prosthesis.

By using a planning program with treatment simulation through the use of our own virtual models for standard prostheses, virtual planning of jaw and prosthesis positioning is possible even with a standardized temporomandibular joint prosthesis. In this way, the advantages of virtual planning are partly brought to the patients at a much lower price.

This project aims to virtually plan treatment for patients with standardized temporomandibular joint prosthesis. Patients eligible for this study are included retrospectively (have already been treated). Their X-rays will be used for treatment planning and for comparison with the treatment outcome of previous TMJ treatment.

The study will analyze the possibilities of the standardized prostheses to provide the same positions, temporomandibular joint replacements and movements of the jaw as an individual temporomandibular joint prosthesis has. This is done by measuring the planned positions of standardized temporomandibular joint prostheses compared to the treatment outcome shown by previous postoperative X-ray examinations.

The study aims to clarify the possibilities of a simpler and less expensive technology, standardized temporomandibular joint prostheses, to achieve the same good treatment outcome as a more costly technology. This with the same possibilities for treatment planning and use that the existing, more expensive technology, individual temporomandibular joint prostheses, has today.

DETAILED DESCRIPTION:
Aim and objectives

The aim of the present study was to evaluate the possibility to perform patient specific treatment planning with the use of standardized total TMJ prosthesis on previously performed treatment with total TMJ replacement and occlusal adjustment due to a severe malocclusion. The objectives were surgical feasibility of virtual planning on standardized TMJ prosthesis measuring virtual possible maximal interface (mm2) between prosthesis and bone, possible maximal number of fixation screws and possibility to centre the mandibular part in the fossa part. The outcome measures were surgical movements to correct a severe malocclusion using standardized TMJ prosthesis.

Survey of the field

A total replacement of the temporomandibular joint (TMJ) has been successfully offered to patients with severe joint disease since more than three decades. In the early years, the surgical technique has been judged as complex and similar to other joint prosthesis the TMJ prosthesis has been burdened with some risk of complications. With emerging technologies, within computer science, biomedical design, and biocompatible materials the treatment option has been possible to use in a wider perspective. Thus, a broader patient spectrum has been possible to rehabilitate with TMJ prosthesis. Today, not only joint-related pathologic conditions are offered joint reconstruction, but also congenital deformities like Hemifacial Microsomia and Dentofacial deformities. Furthermore, the advancement of the treatment quality has enabled patients with severe joint-pathology, like Juvenile Idiopathic Arthrosis with a subsequent severe malocclusion and facial deformity, to have a total rehabilitation with both normalization of the joint function together with improved facial appearance and bite function.

However, in many of these severe cases the corrections of the facial structures simultaneously with a joint replacement provides the surgeon with a complex treatment-planning phase. Frequently, the movements need to be planned and simulated virtually to evaluate both the best positioning of segments and joint components and to manufacture surgical indexes and cutting templates. The invention of patient specific solutions (PSI) have made hardware design based on 3D radiological imaging and soft tissue predictions possible. Patient specific total TMJ prosthesis provided the surgeon with virtual planning, cutting guides, occlusal splints and well-fitted alloplastic TMJ components. However, this came with additional costs and the advantage of customized prosthesis over standardized have been debated. Attempts have been made to retrospectively compare customized with standard prosthesis, but this fare no prospective or RCT have been published. Presently, this lack of prospective comparisons leaves the evaluation with only retrospective and observational comparisons. This results in a risk of bias because of a difference in treatment indication between the compared treatment modalities. Thus, the outcome from a retrospective comparison will be coloured by a selection bias with the indication for treatment as a confounding factor.

However, while most patients with TMD might facilitate by treatment with less invasive methods than TMJ prosthesis, the other patient categories mentioned are not in a situation where they have alternative methods nor having less treatment need within time. Treating such patients at an early stage would give a rehabilitation that address all their treatment goals simultaneously, adding more years to a lifetime, with a normalized condition and a better quality of life. This with the most available and cost-effective method provided, i.e. analysis cost-utility measures using QALY. Today, a more cost-efficient treatment method might be possible using standardized total TMJ replacement prosthesis, with less cost compared with customized, in a customized planning system like VSP orthognathic surgery planning for occlusal adjustment. However, there is a possible limitation for the use of a standardized TMJ prosthesis in those patients where the anatomy of the TMJ and adjacent structures, due to pathology and/or congenital deformities, differ much from ordinary anatomy. This far, there are no clear guidelines to when a standardized TMJ prosthesis is possible to use or when any limitations of its design lead to a need of choosing a customized prosthesis.

Traditional advantages of stock devices include lower cost and immediate availability. Furthermore, stock devices work well in most cases with normal anatomy.30 It has also been stated that custom joints are implanted with a higher level of accuracy due to the feature of a virtual surgical planning (VSP). However, with a possibility to use VSP even for standard TMJ prosthesis, this advantage will no longer advocate the choice of a method that is more time-consuming and to a higher price.

The scientific hypothesis of the present study was that most TMD-caused severe malocclusions treated with a total TMJ replacement, that traditionally would be treated by a PSI TMJ prosthesis, would be possible to perform using virtual surgical planning with a standardized TMJ prosthesis.

Description of the project

Subjects

A retrospective observation study will be performed on patients treated with standard prosthesis in combination with three-dimensional virtual planning. Patients included were treated at the department of Oral and Maxillofacial Surgery, Skåne University Hospital. Lund, Sweden during 2010 to 2024.

Method

Preoperative radiographs will be used for re-evaluation of possibilities for virtual surgical planning on standardized total TMJ reconstruction.

The radiographs will during 2025 be used for a secondary treatment planning with virtual models of standardized TMJ prosthesis. Pre- and post-treatment radiographs will be analyzed, virtually treatment planned and simulated with standard prostheses in a virtual planning program. This secondary and retrospective treatment planning will be performed with the same jaw movements as were previously achieved. Three-dimensional cephalometric measurements of distances and angles between standardized landmarks will be performed in the pre- and postoperative CT images. Changes in landmark positions in the two examinations will be recorded as a measure of surgical differences.

Time plan (preliminary) Project start: 2026-01-01 Project closure: 2027-12-31

Importance

The difference between previously performed treatment and a new virtual planning in this study is that only standard prostheses will be used for temporomandibular joint reconstruction and bite correction. The method that is intended to be tested in this project combines the advantages of virtual planning with the economic advantages of standard design of temporomandibular joint prostheses.

Preliminary results

Today, no studies have been published on the combination of standardized prosthesis design and virtual planning of jaw surgery.

The method of virtual surgical planning, has been used by the applicant for this ethical review for more than 20 years and has been studied in several published clinical trial.

The method, that is intended to be tested in this project, combines the advantages of virtual planning with the economic advantages of standard design of temporomandibular joint prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe pathology in the temporomandibular joint.
* Previously treated with TMJ prosthesis at the department of Oral and Maxillofacial Surgery, Skåne University Hospital, Lund, Sweden.
* Treatments performed during year 2010 to 2025.

Exclusion Criteria:

- Patients with additional surgical treatment of the TMJ after total TMJ replacement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously treated with TMJ prosthesis at the department of Oral and Maxillofacial Surgery, Skåne University Hospital. Lund, Sweden during 2010 to 2025.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurements in preoperative radiographs for re-evaluation of possibilities for virtual surgical planning on standardized total TMJ reconstruction. | During 2026 retrospective virtual measurement on previous radiographs will be performed. Because patient treatments were performed during 2010 to 2025 the measurements will be performed 1 to 16 years after the recordings were performed
  Measurements in images from virtual planned standardized TMJ prosthesis will include the following variables:
  * Maximal interface between bone tissue and prosthesis surface (mm2)
  * Size Fossa component
  * Size Mandibular component
  * Maximal number of fixation screws
  * Centre the mandibular part in the fossa part.
  * Angle between fossa and mandible part (frontal)
  * Angle between fossa and mandible part (sagittal)

SECONDARY OUTCOMES:
Recorded surgical movements to correct a severe malocclusion. | During 2026 retrospective virtual measurement on previous radiographs will be performed. Because patient treatments were performed during 2010 to 2025 the measurements will be performed 1 to 16 years after the recordings were performed.
  Registrations from patient journals and radiographs will include the following variables:
  * Occlusal reposition
  * Maxillary reposition
  * Mandibular movement
  * Size Fossa component
  * Size Mandibular component
  * Use of bone transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Surgery, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 12. Zou L, He D, Ellis E. A Comparison of Clinical Follow-Up of Different Total Temporomandibular Joint Replacement Prostheses: A Systematic Review and Meta-Analysis. J Oral Maxillofac Surg 2018;76:294-303.
- [Background] 11. de Las Fuentes Monreal M, Escorial Hernandez V, Garcia Jimenez T, Munoz-Guerra MF. Revision of the Wolford protocol for managing infections in temporomandibular joint prostheses: an updated surgical approach. Int J Oral Maxillofac Surg 2024;53:1065-1067.
- [Background] 10. Peres Lima FGG, Rios LGC, Bianchi J, Goncalves JR, Paranhos LR, Vieira WA, et al. Complications of total temporomandibular joint replacement: a systematic review and meta-analysis. Int J Oral Maxillofac Surg 2023;52:584-594.
- [Background] 9. Bach E, Sigaux N, Fauvernier M, Cousin AS. Reasons for failure of total temporomandibular joint replacement: a systematic review and meta-analysis. Int J Oral Maxillofac Surg 2022;51:1059-1068.
- [Background] 8. Wolford LM, Pitta MC, Reiche-Fischel O, Franco PF. TMJ Concepts/Techmedica custom-made TMJ total joint prosthesis: 5-year follow-up study. Int J Oral Maxillofac Surg 2003;32:268-274.
- [Background] 7. Rajkumar A, Sidebottom AJ. Prospective study of the long-term outcomes and complications after total temporomandibular joint replacement: analysis at 10 years. Int J Oral Maxillofac Surg 2022;51:665-668.
- [Background] 6. O'Connor RC, Saleem S, Sidebottom AJ. Prospective outcome analysis of total replacement of the temporomandibular joint with the TMJ Concepts system in patients with inflammatory arthritic diseases. Br J Oral Maxillofac Surg 2016;54:604-609.
- [Background] 5. Johnson NR, Roberts MJ, Doi SA, Batstone MD. Total temporomandibular joint replacement prostheses: a systematic review and bias-adjusted meta-analysis. Int J Oral Maxillofac Surg 2017;46:86-92.
- [Background] 4. Ravelo V, Vargas E, Garcia Guevara H, Sacco R, Navarro P, Olate S. TMJ Replacement in Degenerative Disease: A Systematic Review. J Clin Med 2025;14.
- [Background] 3. Lima F, Rios LGC, Paranhos LR, Vieira WA, Zanetta-Barbosa D. Survival of temporomandibular total joint replacement: A systematic review and meta-analysis. Journal of oral rehabilitation 2024;51:775-784.
- [Background] 2. Leandro LF, Ono HY, Loureiro CC, Marinho K, Guevara HA. A ten-year experience and follow-up of three hundred patients fitted with the Biomet/Lorenz Microfixation TMJ replacement system. Int J Oral Maxillofac Surg 2013;42:1007-1013.
- [Background] 1. Giannakopoulos HE, Sinn DP, Quinn PD. Biomet Microfixation Temporomandibular Joint Replacement System: a 3-year follow-up study of patients treated during 1995 to 2005. J Oral Maxillofac Surg 2012;70:787-794; discussion 795-786.